CLINICAL TRIAL: NCT07195227
Title: Phase II Study to Evaluate the Efficacy and Safety of Camizestrant Plus Ribociclib in Patients With Hormone Receptor Positive (HR+) Breast Cancer
Brief Title: Efficacy and Safety of Camizestrant Plus Ribociclib in Patients With Breast Cancer
Acronym: CADILLAC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP555
Record Dates: First submitted 2025-06-10; First posted 2025-09-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hormon Receptor Positive Breast Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A: Camizestrant and Ribociclib (Experimental): Patients will receive Camizestrant (75 mg, oral, every day on each day of the 28-day cycle) and Ribociclib (600 mg, oral, every day, on day 1 to 21 of each 28-day cycle)
  Interventions: Drug: Camizestrant; Drug: Ribociclib
- Control Arm B: Historical Arm (No Intervention): The clinical Study comparator will be a historical control arm containing data from all or some of the following clinical trials: MONALEESA-2, MONALEESA-3, MONALEESA-7, CompLEEment-1, and RIBECCA.

INTERVENTIONS:
Drug: Camizestrant — Next-generation oral SERD molecule that is intended for the treatment of women and men with ER+ breast cancer. In addition to degradation of ERα, camizestrant also acts as a pure ER antagonist
  Arms: Experimental Arm A: Camizestrant and Ribociclib
Drug: Ribociclib — Selective inhibitor of CDK 4 and 6, with 50% inhibition (IC50) values of 0.01 μM (4.3 ng/ml) and 0.039 μM (16.9 ng/ml) in biochemical assays, respectively. These kinases are activated by binding to D-cyclins and are crucial to cell cycle progression and cellular proliferation. The cyclin D-CDK4/6 complex regulates the cell cycle by phosphorylating the retinoblastoma protein (pRb).
  Arms: Experimental Arm A: Camizestrant and Ribociclib

SUMMARY:
This trial will study a type of breast cancer defined by the expression of hormone receptor in the cancer cells (HR+). Patients will be treated with ribociclib, a cyclin-dependent kinase inhibitor, and camizestrant, a selective estrogen receptor degrader (SERD) and complete ER antagonist. The main purpose of the Study is to analyze the efficacy (to find out how effective a treatment is) of ribociclib in combination with camizestrant in patients with advanced HR+ breast cancer who have received endocrine therapy (ET) in early breast cancer setting for at least 5 years, of which at least 2 years with aromatase inhibitor (AI). Ribociclib plus camizestrant efficacy will be determined by assessing the period from treatment initiation until disease progression, defined as progression free survival (PFS).

The anticipated favorable clinical benefits of the combination of ribociclib and camizestrant therapy are projected to outweigh the risks of this treatment. This Study will be performed in full compliance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) and all applicable local Good Clinical Practice (GCP) and regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be capable of understanding the purpose of the Study and have signed the written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female or male patients ≥ 18 years of age at the time of signing ICF.
3. Pre- or peri-menopausal women or men. are eligible if treated with a Luteinizing hormone-releasing hormone (LHRH) analogue. Treatment with a LHRH is recommended for at least 28 days prior to study treatment; if shorter, post-menopausal levels of serum estradiol/follicle-stimulating hormone [FSH] must be confirmed analytically prior to Study enrollment.
4. Post-menopausal women, defined by any of the following criteria:

   * Cessation of menses for at least 12 consecutive months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
   * Documented bilateral surgical oophorectomy.
5. Documented histologically confirmed HR+ and human epidermal growth factor receptor 2 (HER2)-negative breast cancer according to the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines as per local assessment on the most recent analyzed biopsy. Therefore, tumors must be:

   o HR+ defined as ≥ 10% of tumor cells stain positive for estrogen receptor (ER) on immunohistochemistry (IHC), and HER2- defined as 0 or 1+ intensity on IHC, or 2+ intensity on IHC and no evidence of amplification on in situ hybridization (ISH).
6. Unresectable locally recurrent or metastatic disease confirmed by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
7. Patients must have received at least five years of adjuvant endocrine therapy, including at least two years of an AI (capped to 30% patients with treatment-free interval [TFI] ≥ 12 months.
8. Patients must have:

   * Radiological evidence of progression while on, or within 12 months of the end of (neo)adjuvant endocrine therapy (secondary endocrine resistance criteria), or
   * Radiological evidence of progression more than 12 months of the end of (neo)adjuvant endocrine therapy (endocrine sensitive criteria).
9. Patients receiving a CDK4/6 inhibitor-based therapy in the (neo)adjuvant setting are eligible if disease progression is confirmed more than 12 months following CDK4/6 inhibitor treatment completion in this scenario.
10. Evidence of measurable disease as per RECIST v.1.1, or non-measurable, but evaluable, disease, including bone-only disease with at least one lytic or mixed lytic-blastic bone lesion.
11. For patients receiving tamoxifen or toremifene, a washout period of 35 days (5 half-lives) prior to randomization is required
12. Patients must agree to provide and have available a FFPE tissue biopsy sample taken at the time of presentation with recurrent or metastatic disease. If this is not available, archived primary breast cancer specimen may be submitted
13. Adequate bone marrow and organ function:

    * Hematological (without platelet, red blood cell transfusion, and/or granulocyte colony-stimulating factor support within seven days before treatment initiation): White blood cell (WBC) count > 3.0 x 109/L; absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 100.0 x109/L; and hemoglobin ≥ 9.0 g/dL.
    * Hepatic: Serum albumin ≥ 2.5 g/dL; total serum bilirubin < 1.5 x upper limit of normal (ULN) except for patients with Gilbert's syndrome who may be included if the total serum bilirubin is ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN; alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 3 x ULN in patients with liver and/or bone metastases); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 x ULN (≤ 3 x ULN in patients with liver metastases); international normalized ratio (INR) < 1.5. Prothrombin time (PT) or Prothrombin time-international normalized ratio (PT-INR) and activated partial thromboplastin time (aPTT)/partial thromboplastin time (PTT) ≤ 1.5 × ULN, except for subjects receiving coumarin-derivative anticoagulants, factor Xa inhibitors, or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator from product safety requirements (PSR).
    * Renal: Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min as calculated by Cockcroft- Gault equation.
14. Patient must be available and willing to participate in the treatment and follow-up assessments as required.
15. Women of childbearing potential who are sexually active with a non-sterilized male partner must have a negative serum pregnancy test within 14 days before Study treatment initiation. In addition, they must agree to use one highly effective method of birth control from the time of screening until 4 weeks after the last dose of Study treatments. Female patients must refrain from egg cell donation and breastfeeding during this same period. Non-sterilized male partners of heterosexually active females of childbearing potential participants must use a male condom from the time of enrollment of their female partner, throughout their participation in the Study, and until 4 weeks after their female partner's last dose of Study intervention.
16. Male participants who are sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable highly effective method of contraception from the time of screening until 21 days after the last administration of the Study drug. Male participants must not donate or bank sperm during this same period. Female partners of childbearing potential of male participants must agree to use one highly effective method of contraception from the time of screening until 4 weeks after the last dose of Study treatments.
17. ECOG performance status of 0-1.
18. Minimum life expectancy of ≥ 6 months.

Exclusion Criteria:

1. Formal contraindication to endocrine therapy defined as visceral crisis and/or rapidly or symptomatic progressive visceral disease.
2. Current participation in another therapeutic clinical trial.
3. Has previously been treated with any SERD, including camizestrant, experimental ETs or fulvestrant.
4. Prior systemic therapy for advanced disease.
5. Known active uncontrolled or symptomatic central nervous system (CNS) metastases and/or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases are eligible if they have been previously treated with local therapy, are clinically stable, and off anticonvulsants and steroids for at least 14 days before the first dose of Study treatment.
6. History of another primary malignancy except for the following:

   1. Malignancy treated with curative intent with no known active disease ≥ 3 years before the first dose of Study treatment, and of very low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease.
   3. Other exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin.

   Note: For other cancers considered to have a low risk of recurrence, discussion with the Medical Monitor is required.
7. Known allergy or hypersensitivity reaction to any investigational medicinal products (IMPs) or their incorporated substances.

   Note: Ribociclib is contraindicated for patients with hypersensitivity/allergy to peanut or soya.
8. History of malabsorption syndrome or other condition that would interfere with enteral absorption (ongoing gastrointestinal obstruction/motility disorder, malabsorption syndrome, or prior gastric bypass) or results in the inability or unwillingness to swallow pills.
9. Palliative radiotherapy with a limited field of radiation within two weeks or with wide field of radiation or radiation to more than 30% of the bone marrow within four weeks prior to Study enrollment.
10. Major surgical procedure or significant traumatic injury within 14 days before Study enrollment.
11. Known abnormalities in coagulation such as bleeding diathesis, or any history of coagulopathy within six months before Study enrollment, including history of deep vein thrombosis or pulmonary embolism.
12. Pregnant or lactating women or patients not willing to apply highly effective contraception as defined in the protocol.
13. Current known infection with human immunodeficiency virus (HIV) detectable viral load, hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
14. Any other active uncontrolled infection at the time of screening. Known substance abuse or any other concurrent severe and/or uncontrolled psychiatric or medical condition that would, in the Investigator's judgment, contraindicate patient participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 28 months
  PFS, defined as the time from the date of the first dose until the first occurrence of disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 28 months
  ORR, defined as the rate of patients with a Best Overall Response (BOR) of complete response or partial response, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1.
Clinical Benefit Rate (CBR) | up to 28 months
  CBR, defined as the rate of patients with objective response (complete or partial response), or stable disease for at least 24 weeks, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1.
Time to Response (TTR) | Up to 28 months
  TTR, defined as the time from the date of the first dose until the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a complete or partial response, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1.
Duration of Response (DoR) | Up to 28 months
  DoR, defined as the period from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1.
Best percentage of change | Up to 28 months
  Best percentage of change from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease will be observed, as determined locally by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1.
Time To Subsequent Line of Chemotherapy (TTSLC) | Up to 28 months
  TTSLC, defined as the time from the date of the first dose until the subsequent line of chemotherapy as determined locally by the investigator.
Patient quality of life assessments | Up to 28 months
  Changes from baseline in the European Organisation for Research and Treatment of Cancer quality of life (QLQ-C30) questionnaire.
Number of patients reporting adverse events | Up to 28 months
  Safety and tolerability, assessed by Adverse Events, Treatment Emergent Adverse Events and Serious Adverse Events incidence (graded according to Common Terminology Criteria for Adverse Events (NCI-CTCAE v.5.0)), dose modifications, clinical laboratory parameters, performance status, and vital signs.
Patient reported quality of life assessments | Up to 28 months
  Changes from baseline in the breast cancer-specific (QLQ-BR42) questionnaire.

IPD SHARING:
Plan to Share IPD: No